CLINICAL TRIAL: NCT07340645
Title: Effect of Acupressure on Anxiety, Embarrassment, and Procedure-Related Fear in Patients Undergoing Urodynamic Testing: A Randomized Controlled Trial
Brief Title: Effect of Acupressure on Anxiety, Embarrassment, and Procedure-Related Fear Undergoing Urodynamic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Dr, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TU-BOZKUL-014
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Anxiety; Embrassment; Fear; Urodynamics
Keywords: urodynamics; fear; Embrassment; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-arm (1:1), randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: During the data collection process, when patients present to the urology outpatient clinic, their eligibility for inclusion in the study will be assessed by the researcher M.B. To eliminate selection bias, block randomization will be applied. Participants will be assigned to the acupressure or control group according to permutations (e.g., ABBAAB, BABABA, etc.) in a randomization list generated by an independent biostatistician using a computer-based program.
  After the randomization list is created, the assignment of groups A and B to either the intervention or control group will be determined by a lottery method. Subsequently, M.B., who will not be involved in the data collection process, will prepare sealed envelopes numbered from 1 to 68 corresponding to the sample size, each containing a letter (A or B) representing the group allocation. M.B. will open the numbered envelope and inform GB of the patient's group assignment.
  All researchers other than M.B. will be blinded to the gro
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Acupressure group (Experimental): The acupressure points to be used include Shen Men (HT7), located in the small depression between the pisiform and ulna bones at the transverse wrist crease; EX-NH3, located at the midpoint between the eyebrows on the midline of the forehead; and Hegu (LI4), located in the web space between the thumb and index finger. These points will be marked with an acetate pen on patients in the intervention group by a certified researcher (GB), and the acupressure application will also be performed by the same certified researcher (GB). Patients in the control group will not receive any intervention and will receive routine care only.
  Interventions: Other: Acupressure
- Control group (No Intervention): The control group will receive routine care.

INTERVENTIONS:
Other: Acupressure — The acupressure points to be used include Shen Men (HT7), located in the small depression between the pisiform and ulna bones at the transverse wrist crease; EX-NH3, located at the midpoint between the eyebrows on the midline of the forehead; and Hegu (LI4), located in the web space between the thumb and index finger. These points will be marked with an acetate pen on patients in the intervention group by a certified researcher (GB), and the acupressure application will also be performed by the same certified researcher (GB). Patients in the control group will not receive any intervention and will receive routine care only.
  Arms: Experimental: Acupressure group

SUMMARY:
The study was planned as a randomized controlled experimental design to determine the effect of acupressure on anxiety, embarrassment, and procedure-related fear in patients undergoing urodynamic testing. Since no similar study was identified in the literature for sample size calculation, an effect size of 0.8, which is considered a large effect, was taken as a reference. With 90% power (1-α, two-tailed), the minimum required sample size was calculated using the G*Power (version 3.1) program as 68 participants, with 34 individuals in each group (intervention group = 34; control group = 34). A post hoc power analysis will also be conducted.

Data will be collected using a Sociodemographic Information Form, the Embarrassment Assessment Scale, the State Anxiety Inventory, and the Procedure-Related Fear Scale. Individuals included in the sample will be informed about the study and the procedures to be followed, and their verbal and written informed consent will be obtained. All patients will complete the Sociodemographic Information Form, the Embarrassment Assessment Scale, the State Anxiety Inventory, and the Procedure-Related Fear Scale. After the forms are completed and recorded, participants will be assigned to either the intervention or control group according to the randomization schedule.

In the intervention group, acupressure will be performed by a certified researcher (GB) who has completed acupressure training. The acupressure points to be used include Shen Men (HT7), located in the small depression between the pisiform and ulna bones on the transverse wrist crease; EX-NH3, located at the midpoint between the eyebrows on the midline of the forehead; and Hegu (LI4), located in the web space between the thumb and index finger. These points will be marked with an acetate pen by the certified researcher (GB) in patients assigned to the intervention group, and the application will be carried out by the same researcher.

No intervention will be applied to patients in the control group, and they will receive routine care only.

All patients in both the intervention and control groups will complete the Embarrassment Assessment Scale, the State Anxiety Inventory, and the Procedure-Related Fear Scale. After completion of the acupressure application, the urodynamic procedure will be performed. Immediately after the procedure, patients in both groups will again complete the Embarrassment Assessment Scale, the State Anxiety Inventory, and the Procedure-Related Fear Scale.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled experimental design to determine the effect of acupressure on anxiety, embarrassment, and procedure-related fear in patients undergoing urodynamic testing. Since no similar study was identified in the literature for sample size calculation, an effect size of 0.8, which is considered a large effect, was taken as a reference. With 90% power (1-α, two-tailed), the minimum required sample size was calculated using the G*Power (version 3.1) program as 68 participants, with 34 individuals in each group (intervention group = 34; control group = 34). A post hoc power analysis will also be conducted.

Data will be collected using a Sociodemographic Information Form, the Embarrassment Assessment Scale, the State Anxiety Inventory, and the Procedure-Related Fear Scale. Individuals included in the sample will be informed about the study and the procedures to be followed, and their verbal and written informed consent will be obtained. All patients will complete the Sociodemographic Information Form, the Embarrassment Assessment Scale, the State Anxiety Inventory, and the Procedure-Related Fear Scale. After the forms are completed and recorded, participants will be assigned to either the intervention or control group according to the randomization schedule.

In the intervention group, acupressure will be performed by a certified researcher (GB) who has completed acupressure training. The acupressure points to be used include Shen Men (HT7), located in the small depression between the pisiform and ulna bones on the transverse wrist crease; EX-NH3, located at the midpoint between the eyebrows on the midline of the forehead; and Hegu (LI4), located in the web space between the thumb and index finger. These points will be marked with an acetate pen by the certified researcher (GB) in patients assigned to the intervention group, and the application will be carried out by the same researcher.

No intervention will be applied to patients in the control group, and they will receive routine care only. Before starting the application in the intervention group, the tissue around the marked points will be gently rubbed to promote relaxation. Pressure will then be applied to the marked points using the index or middle finger, creating a depth of approximately 1-1.5 cm for 5 seconds, followed by a 2-second rest. Each point will be stimulated for 3 minutes, with the total duration of the application lasting approximately 15-20 minutes.

All patients in both the intervention and control groups will complete the Embarrassment Assessment Scale, the State Anxiety Inventory, and the Procedure-Related Fear Scale. After completion of the acupressure application, the urodynamic procedure will be performed. Immediately after the procedure, patients in both groups will again complete the Embarrassment Assessment Scale, the State Anxiety Inventory, and the Procedure-Related Fear Scale.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the study,
* 18 years of age or older,
* Conscious, oriented and cooperative,
* No communication problems,
* Individuals undergoing invasive urodynamic procedures.

Exclusion Criteria:

* Who did not agree to participate in the study,
* Under 18,
* Conscious, oriented and uncooperative,
* Communication problems,
* Individuals who did not undergo invasive urodynamics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Embrassment | 10 months
  To assess the level of embrassment, the Visual Analog Scale (VAS) will be used. The scale allows for the subjective evaluation of embrassment on a horizontal or vertical line ranging from 0 (not afraid at all) to 10 (extremely afraid).
Anxiety | 11 months
  The State Anxiety Scale : The DAQ consists of 20 questions on a four-point Likert scale. The statements in the DAQ are evaluated as not at all (1), a little (2), a lot (3) and completely (4). In this section, the statements are divided into direct and reversed statements. Inverted statements: 1st, 2nd, 5th, 5th, 8th, 8th, 10th, 11th, 15th, 16th, 19th, 20th items. The total score of the reversed statements is subtracted from the total score of the direct statements and the number 50, which is the invariant value of the DAQ, is added to the value obtained and the DAQ score is calculated. The scale score ranges between 20-80 and an increase in the score indicates an increase in the level of anxiety.
Fear | 10 months
  To assess the level of procedure-related fear, the Visual Analog Scale (VAS) will be used. The scale allows for the subjective evaluation of procedure-related fear on a horizontal or vertical line ranging from 0 (not afraid at all) to 10 (extremely afraid).

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Bozkul, Study Chair — Tarsus University; Gülay Altun Uğraş, Principal Investigator — Mersin University; MURAT BOZLU, Principal Investigator — Mersin University; ELİFE KETTAŞ DÖLEK, Principal Investigator — Mersin University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozturk E, Hamidi N, Yikilmaz TN, Ozcan C, Basar H. Effect of Listening to Music on Patient Anxiety and Pain Perception during Urodynamic Study: Randomized Controlled Trial. Low Urin Tract Symptoms. 2019 Jan;11(1):39-42. doi: 10.1111/luts.12191. Epub 2017 Aug 23. PMID 28834330
- [Background] Kettas Dolek E, Altun Ugras G. The effect of aromatherapy during urodynamic testing on patients anxiety and cortisol levels: A randomized controlled trial. Neurourol Urodyn. 2024 Sep;43(7):1591-1599. doi: 10.1002/nau.25491. Epub 2024 May 15. PMID 38747020
- [Background] Jiang ZF, Liu G, Sun XX, Zhi N, Li XM, Sun R, Zhang H. Auricular acupressure for constipation in adults: a systematic review and meta-analysis. Front Physiol. 2023 Oct 16;14:1257660. doi: 10.3389/fphys.2023.1257660. eCollection 2023. PMID 37908337
- [Background] Drake MJ, Doumouchtsis SK, Hashim H, Gammie A. Fundamentals of urodynamic practice, based on International Continence Society good urodynamic practices recommendations. Neurourol Urodyn. 2018 Aug;37(S6):S50-S60. doi: 10.1002/nau.23773. PMID 30614058
- [Background] Chen YW, Wang HH. The effectiveness of acupressure on relieving pain: a systematic review. Pain Manag Nurs. 2014 Jun;15(2):539-50. doi: 10.1016/j.pmn.2012.12.005. Epub 2013 Feb 15. PMID 23415783
- [Background] Biardeau X, Lam O, Ba V, Campeau L, Corcos J. Prospective evaluation of anxiety, pain, and embarrassment associated with cystoscopy and urodynamic testing in clinical practice. Can Urol Assoc J. 2017 Mar-Apr;11(3-4):104-110. doi: 10.5489/cuaj.4127. PMID 28515809